CLINICAL TRIAL: NCT05086926
Title: Feasibility of a Home Exercise Program With the Addition of a Corticosteroid Injection in Patients With Greater Trochanteric Pain Syndrome in General Practice
Brief Title: Feasibility of Home Exercises With the Addition of a Corticosteroid Injection in Patients With Lateral Hip Pain in General Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Sabina Vistrup, MD, PhD student, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Study3-2021
Record Dates: First submitted 2021-09-14; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Lateral Hip Pain; Gluteal Tendinopathy; Greater Trochanteric Pain Syndrome
MeSH Terms: interventions — Exercise; Craniospinal Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercises and CSI (Experimental): A corticosteroid injection in the lateral hip prior to performing an 8-week home exercise program
  Interventions: Combination Product: Exercises and CSI

INTERVENTIONS:
Combination Product: Exercises and CSI — Corticosteroid injection:
  The project manager will give the participants one injection with cortisone and lidocaine in the lateral hip at baseline. The procedure will be performed aseptically.
  Home exercise program:
  The exercise programis based on previous literature and expert opinions that has been synthesized in a Delphi study conducted by our research group. The exercise program consists of three body weighted strength exercises, that are to be performed every second day for a period of 8 weeks. Exercise instructions will be available as a handout and online with video instructions. The corticosteroid injection usually causes a flare-up in pain with a duration of up to 48 hours. Participants will be instructed to begin the exercises as soon as possible after this flare-up has settled.

SUMMARY:
Pain on the lateral side of the hip is a common condition in general practice, however there is limited evidence on how to best manage the condition. The purpose of this study is to evaluate the feasibility of a combined treatment before comparing this treatment in a larger clinical trial. For the present study 20 patients with lateral hip pain will be invited to receive a corticosteroid injection in the lateral hip prior to performing our exercise program for 8 weeks. After 4 weeks we will do a short interview to get feedback on the exercise program. After 8 weeks we will evaluate the acceptability of the combined treament.

DETAILED DESCRIPTION:
BACKGROUND:

Lateral hip pain or greater trochanteric pain syndrome (GTPS) is pain on the outside of the hip due to tendon pathology of the hip abductor tendons. The incidence in primary care has been reported to be 1.6-3.3 per 1000 patients per year. At present, there is no evidence-based guidelines for the treatment of GTPS in primary care. The investigators of the present study have developed an exercise protocol that is planned be evaluated in a future randomized controlled trial in combination with a corticosteroid injection.

OBJECTIVE:

The purpose of this study is to evaluate feasibility of a home exercise program with the addition of a corticosteroid injection in patients with GTPS in general practice. The primary aim is to evaluate patient acceptability of 1) performing our exercise program 2) performing exercises after receiving a corticosteroid injection. The secondary aim is to obtain feedback from patients through qualitative interviews to be able to refine the exercise intervention after the study is completed. If the combined treatment is found feasible, it is planned to evaluate the effect in a large randomized controlled trial in the future.

STUDY DESIGN:

The study design is a mixed methods feasibility study. The participants are patients with GTPS that will receive a combined treatment of one corticosteroid injection in the lateral hip and a home exercise program, which is to be performed for a period of eight weeks. The acceptability of the combined intervention will be evaluated after 8 weeks.

RECRUITMENT OF PARTICIPANTS:

Patients with GTPS will be recruited from general practice and a private rheumatology practice. Patients will be considered for inclusion if they present to their practitioner with self-reported lateral hip pain. The project manager will make a screening of eligibility by telephone. Those not excluded based on this screening, will be invited to a clinical examination where final eligibility is determined.

ENDPOINTS:

Baseline is at the clinical examination. One week from baseline there will be a short phone contact to the participants in order to clarify any questions related to the exercise program. No data will be obtained at this point. At 4 weeks there will be a phone interview which also serves as a booster session where the participants are encouraged to maintain their exercise routine. At 8 weeks there will be a physical visit where the participants will hand in their exercise diaries and complete the final questionnaires.

CRITERIA OF FEASIBILITY:

To conclude that the combined treatments are feasible, ≥ 75% of patients must rate the treatment as 'acceptable'. If any participant drops out after the injection, they will be dichotomized as "not acceptable". A minimum of 15/20 training diaries must be handed in at 8-weeks follow-up. Based on the returned training diaries, ≥ 75% of participants need to complete ≥ 20/28 possible training sessions. A training session will be considered completed if the participant has performed at least one set of each exercise.

In case the combined treatments do not prove feasible according to this set of criteria, it is planned to refine the intervention based on feedback from the interviews and evaluate with a small group of patients for a shorter period of time.

ELIGIBILITY:
Inclusion Criteria:

* >35 years of age
* Self-reported pain on the outside of the hip for at least 12 weeks with an average intensity of present pain over the last week of at least 4/10 on a numeric rating scale 0-10 (0 being no hip pain and 10 being worst hip pain imaginable)
* Access to a computer, smartphone or tablet with internet connection
* Tenderness on palpation of the greater trochanter
* Reproduction of lateral hip pain with 30 sec single leg stance test
* Ability to speak and understand Danish (written and oral)
* In case of bilateral hip pain, the study hip will be the most painful at inclusion

Exclusion Criteria:

* Corticosteroid injection in the affected hip or other new treatment by a health professional within the last 3 months
* History of systemic inflammatory diseases, e.g. rheumatoid arthritis, spondyloarthritis
* Weekly intake of oral glucocorticoids
* History of other hip conditions, e.g. clinically significant hip osteoarthritis, hip dysplasia, prior hip surgery
* History of prior lumbar back surgery
* Current low back pain or episodes of low back pain within the last 3 months that have caused sick leave and/or treatment by a health professional
* Physical or mental disabilities that make it impossible to understand and/or perform exercises and complete questionnaires
* Current or planned pregnancy or breastfeeding

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Acceptability of performing our exercise program | 8 weeks
  7-point Likert scale range "very unacceptable" to "very acceptable"
Acceptability of performing exercises after receiving a corticosteroid injection | 8 weeks
  7-point Likert scale range "very unacceptable" to "very acceptable"

SECONDARY OUTCOMES:
Global Rating of Change | 4 and 8 weeks
  This is determined by asking the question "How is your lateral hip pain now compared to when you first came in for treatment in this project?", which will be responded to with a 7-point Likert scale ranging from "very much worse" to "very much better".
Patent Acceptable Symptom State | 4 and 8 weeks
  This will be identified by asking the patient to answer yes or no to the question "Is your lateral hip pain at an acceptable level that does not require any further treatment?"
Pain Self-Efficacy Questionnaire | 4 and 8 weeks
  This is a self-reported measure used to assess how confident patients are in performing activities while in pain. The outcome is a score of 0 to 60, with higher score indicating higher self-efficacy. We will use a Danish validated version
Health-related quality of life | 4 and 8 weeks
  We will use EuroQol-5D-5L. This is a standardized instrument to assess health related quality of life.
Compliance to exercises | 8 weeks
  Participants will record their exercise sessions using an exercise diary

OTHER OUTCOMES:
Qualitative outcomes | 4 weeks
  Short interview to obtain qualitative feedback from participants. Questions:
  How was your experience in general with completing this exercise program? Which challenges did you experience? How did you find the difficulty of the levels in the exercise program? Did you have any challenges with the training diary? Did you find the phone call from the project manager at one week useful?

CONTACTS AND LOCATIONS:
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No